CLINICAL TRIAL: NCT05286450
Title: Non-compliance on Treatment Among Diabetic Students at Sohag University
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Samah Wagdy Abdelaziz, Demonstrator at Family Medicine Department, Sohag University
Other Study IDs: Soh-Med-22-03-14
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study on diabetic students in Sohag University will be conducted to collect data about factors affecting compliance and adherence to diabetes treatment and its impact on development of complications.

DETAILED DESCRIPTION:
Personal interviews with diabetic students through a questionnaire :

1. To determine factors affecting non compliance on treatment among diabetic students.
2. To detect relation between non compliance on treatment and development of complications.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic students at Sohag University age from 17 to 25

Exclusion Criteria:

* Healthy students
* Students in other universities

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all the diabetic students in sohag university from different faculties
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samah W. Elkhayat, demonstrator, Principal Investigator — Faculty of Medicine Sohag University
Locations (1):
- Faculty of medicine Sohag University, Sohag, Egypt

RESULTS

PARTICIPANT FLOW:
Groups:
- Diabetic Students at Sohag University: 153 diabetic students aged between 17 and 25 years old in different faculties in Sohag University
Period: Overall Study
Arm/Group | Diabetic Students at Sohag University
Started | 153
Completed | 153
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Diabetic Students at Sohag University
Number analyzed (Participants) | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 153
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 153

OUTCOME MEASURES:

1. Primary Outcome: Distribution of Participants Responses as Regards DSMQ Glucose Management Domain
Description: through a standardized questionnaire DSMQ (Diabetes self management questionnaire)
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- Diabetic Students at Sohag University: 153 diabetic students aged between 18 and 25 years old in different faculties in Sohag University
Arm/Group | Diabetic Students at Sohag University
Number analyzed (Participants) | 153
Participants
  I check my blood sugar levels with care and attention.: Does not apply to me | 13
  I check my blood sugar levels with care and attention.: Applies to me to some degree | 56
  I check my blood sugar levels with care and attention.: Applies to me to a consider-able degree | 39
  I check my blood sugar levels with care and attention.: Applies to me very much | 45
  I take my diabetes medication (e. g. insulin, tablets) as prescribed: Does not apply to me | 1
  I take my diabetes medication (e. g. insulin, tablets) as prescribed: Applies to me to some degree | 12
  I take my diabetes medication (e. g. insulin, tablets) as prescribed: Applies to me to a consider-able degree | 32
  I take my diabetes medication (e. g. insulin, tablets) as prescribed: Applies to me very much | 108
  I record my blood sugar levels regularly (or analyse the value chart with my blood glucose meter).: Does not apply to me | 20
  I record my blood sugar levels regularly (or analyse the value chart with my blood glucose meter).: Applies to me to some degree | 51
  I record my blood sugar levels regularly (or analyse the value chart with my blood glucose meter).: Applies to me to a consider-able degree | 35
  I record my blood sugar levels regularly (or analyse the value chart with my blood glucose meter).: Applies to me very much | 47
  I do not check my blood sugar levels frequently as required for achieving good blood glucose control: Does not apply to me | 61
  I do not check my blood sugar levels frequently as required for achieving good blood glucose control: Applies to me to some degree | 37
  I do not check my blood sugar levels frequently as required for achieving good blood glucose control: Applies to me to a consider-able degree | 39
  I do not check my blood sugar levels frequently as required for achieving good blood glucose control: Applies to me very much | 16
  I tend to forget to take or skip my diabetes medication (e. g. insulin, tablets).: Does not apply to me | 120
  I tend to forget to take or skip my diabetes medication (e. g. insulin, tablets).: Applies to me to some degree | 23
  I tend to forget to take or skip my diabetes medication (e. g. insulin, tablets).: Applies to me to a consider-able degree | 7
  I tend to forget to take or skip my diabetes medication (e. g. insulin, tablets).: Applies to me very much | 3

2. Primary Outcome: Distribution of Participants Responses as Regards DSMQ Dietary Control Domain
Description: non compliance on treatment among diabetic students
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Students at Sohag University
Number analyzed (Participants) | 153
Participants
  The food I choose to eat makes it easy to achieve optimal blood sugar levels.: Does not apply to me | 12
  The food I choose to eat makes it easy to achieve optimal blood sugar levels.: Applies to me to some degree | 71
  The food I choose to eat makes it easy to achieve optimal blood sugar levels.: Applies to me to a consider-able degree | 43
  The food I choose to eat makes it easy to achieve optimal blood sugar levels.: Applies to me very much | 27
  Occasionally I eat lots of sweets or other foods rich in carbohydrates: Does not apply to me | 33
  Occasionally I eat lots of sweets or other foods rich in carbohydrates: Applies to me to some degree | 52
  Occasionally I eat lots of sweets or other foods rich in carbohydrates: Applies to me to a consider-able degree | 50
  Occasionally I eat lots of sweets or other foods rich in carbohydrates: Applies to me very much | 18
  I strictly follow the dietary recommendations given by my doctor or diabetes specialist.: Does not apply to me | 30
  I strictly follow the dietary recommendations given by my doctor or diabetes specialist.: Applies to me to some degree | 64
  I strictly follow the dietary recommendations given by my doctor or diabetes specialist.: Applies to me to a consider-able degree | 33
  I strictly follow the dietary recommendations given by my doctor or diabetes specialist.: Applies to me very much | 26
  Sometimes I have real 'food binges' (not triggered by hypoglycemia).: Does not apply to me | 50
  Sometimes I have real 'food binges' (not triggered by hypoglycemia).: Applies to me to some degree | 43
  Sometimes I have real 'food binges' (not triggered by hypoglycemia).: Applies to me to a consider-able degree | 39
  Sometimes I have real 'food binges' (not triggered by hypoglycemia).: Applies to me very much | 21

3. Primary Outcome: Distribution of Participants Responses as Regards DSMQ Physical Activity Domain
Description: mesurment of non compliance among diabetic students at sohag university
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Students at Sohag University
Number analyzed (Participants) | 153
Participants
  I do regular physical activity to achieve optimal blood sugar levels.: Does not apply to me | 90
  I do regular physical activity to achieve optimal blood sugar levels.: Applies to me to some degree | 31
  I do regular physical activity to achieve optimal blood sugar levels.: Applies to me to a consider-able degree | 18
  I do regular physical activity to achieve optimal blood sugar levels.: Applies to me very much | 14
  I avoid physical activity, although it would improve my diabetes.: Does not apply to me | 42
  I avoid physical activity, although it would improve my diabetes.: Applies to me to some degree | 45
  I avoid physical activity, although it would improve my diabetes.: Applies to me to a consider-able degree | 14
  I avoid physical activity, although it would improve my diabetes.: Applies to me very much | 52
  I tend to skip planned physical activity.: Does not apply to me | 37
  I tend to skip planned physical activity.: Applies to me to some degree | 30
  I tend to skip planned physical activity.: Applies to me to a consider-able degree | 25
  I tend to skip planned physical activity.: Applies to me very much | 61

4. Primary Outcome: Distribution of Participants Responses as Regards DSMQ Health Care Use Domain
Description: measurment of non compliance among diabetic students at sohag university
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Students at Sohag University
Number analyzed (Participants) | 153
Participants
  I keep all doctors' appointments recommended for my diabetes treatment: Does not apply to me | 40
  I keep all doctors' appointments recommended for my diabetes treatment: Applies to me to some degree | 60
  I keep all doctors' appointments recommended for my diabetes treatment: Applies to me to a consider-able degree | 26
  I keep all doctors' appointments recommended for my diabetes treatment: Applies to me very much | 27
  I tend to avoid diabetes-related doctors' appointments: Does not apply to me | 72
  I tend to avoid diabetes-related doctors' appointments: Applies to me to some degree | 46
  I tend to avoid diabetes-related doctors' appointments: Applies to me to a consider-able degree | 23
  I tend to avoid diabetes-related doctors' appointments: Applies to me very much | 12
  Regarding my diabetes care, I should see my medical practitioner(s) more often.: Does not apply to me | 46
  Regarding my diabetes care, I should see my medical practitioner(s) more often.: Applies to me to some degree | 49
  Regarding my diabetes care, I should see my medical practitioner(s) more often.: Applies to me to a consider-able degree | 38
  Regarding my diabetes care, I should see my medical practitioner(s) more often.: Applies to me very much | 20
  My diabetes self-care is poor: Does not apply to me | 46
  My diabetes self-care is poor: Applies to me to some degree | 49
  My diabetes self-care is poor: Applies to me to a consider-able degree | 38
  My diabetes self-care is poor: Applies to me very much | 20

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Diabetic Students at Sohag University
All-Cause Mortality (participants affected / at risk) | 0/153
Serious Adverse Events (participants affected / at risk) | 0/153
Other Adverse Events (participants affected / at risk) | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT05286450/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT05286450/SAP_001.pdf